CLINICAL TRIAL: NCT07338227
Title: Validation of Clara Cell Protein as a Novel Diagnostic Biomarker for the Differentiation of Cardiogenic Pulmonary Edema From Non-Cardiogenic Pulmonary Edema
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Foad Ali, Beni Suef general hospital, Egypt., Beni-Suef University
Other Study IDs: 13/3/2024
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Clara Cell Protein; Diagnostic Biomarker; Differentiation; Cardiogenic Pulmonary Edema; Non-Cardiogenic Pulmonary Edema
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPE group: Patients with cardiogenic pulmonary edema
  Interventions: Other: Clara cell protein 16
- NCPE group: Patients with non-cardiogenic pulmonary edema.
  Interventions: Other: Clara cell protein 16

INTERVENTIONS:
Other: Clara cell protein 16 — Clara cell protein 16 (CC16) concentration was measured in serum samples drawn within 24 hours of intubation.

SUMMARY:
This study aimed to validate the use of clara cell secretory protein (CC16) as a biomarker for differentiating between cardiogenic pulmonary edema (CPE) and non-cardiogenic pulmonary edema (NCPE).

DETAILED DESCRIPTION:
Club cells or Clara cells (CCs) were first described in 1881 but their importance was forgotten until Max Clara's 1937 study identifying these bronchiolar exocrine cells. CCs constitute up to 44% of proliferating small airway cells, functioning as epithelial progenitors during lung regeneration and repair of injury.

CC16 can be useful in distinguishing between cardiogenic pulmonary edema (CPE), caused by increased pressure in the heart's left ventricle, and non-cardiogenic pulmonary edema, such as acute lung injury (ALI) or acute respiratory distress syndrome (ARDS), which are not related to heart failure. Patients with ALI/ARDS tend to have lower levels of CC16 in their plasma and pulmonary edema fluid compared to those with CPE, suggesting a potential diagnostic role for CC16 in these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Both sexes.
* Patients requiring intensive care unit (ICU) admission and intubation.
* Inclusion criteria followed the American-European Consensus Conference diagnostic guidelines for acute lung injury (ALI) and acute respiratory distress syndrome (ARDS): acute respiratory failure onset, bilateral infiltrates on chest radiography, a PaO2/FiO2 ratio below 300 for ALI or 200 for ARDS and no evidence of left atrial hypertension

Exclusion Criteria:

* Critically ill but not intubated.
* Had a mixed cause of pulmonary edema like pneumonia with heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study employed a prospective observational design to evaluate 100 patients receiving intubation, mechanical ventilation, and admission to the critical care department at Beni-Suef General Hospital between January 2023 and January 2024 for cardiogenic or non-cardiogenic pulmonary edema. Ethical approval was obtained from Cairo University's Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Clara cell secretory protein (CC16) level | Within 24 hours of intubation
  Clara cell secretory protein (CC16) level was measured in serum samples drawn within 24 hours of intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.